CLINICAL TRIAL: NCT01455116
Title: Randomized Trial to Determine Whether Mild Induced Hypothermia Can Reduce Mortality in Adult Patients With Septic Shock
Brief Title: The Cooling And Surviving Septic Shock Study (CASS)
Acronym: CASS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Danish Procalcitonin Study Group (Other)
Collaborators: TRYG Foundation (Other); Lundbeck Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-A-2008-086
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Septic Shock
Keywords: Sepsis; Multi organ dysfunction syndrome; Mild Induced Hypothermia
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Hypothermia, Induced; Cool-Down Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild induced hypothermia (Experimental): Induced hypothermia to 32-34 degrees Celsius (90 - 93 degrees Fahrenheit)
  Interventions: Procedure: Mild Induced Hypothermia
- Fever Respect (No Intervention): Standard of care septic shock therapy according to Surviving Sepsis Campaign guidelines

INTERVENTIONS:
Procedure: Mild Induced Hypothermia — Induction of hypothermia to a target temperature of 32 - 34 degrees Celsius (90 - 93 degrees Fahrenheit
  Other Names: Cooling
  Arms: Mild induced hypothermia

SUMMARY:
Septic shock is in critically ill patients is a condition associated with a high rate of organ failure and hereto attributable mortality ~45-55% Hypothesis: Mild Induced Hypothermia reduces the mortality of critically ill patients with septic shock by reducing organ metabolism, counteracting on microcirculatory thrombosis, genetically downregulating tissue apoptosis and by reducing bacterial growth rate and toxin production.

DETAILED DESCRIPTION:
Septic shock is an acute life-threatening condition, with great organ damage for every hour. The patients have a high risk of dying and therefore rapid treatment is of crucial importance for survival of the patients.

Septic shock is mainly due to a collapse in the blood circulation (the capillary system) due to blockage by blood cells - a process initiated by substances from the cells of the immune system via activation of coagulation. The normal function of the smallest blood vessels is to transport oxygen, nutrients and drugs to organs and tissues, and lead waste products away. While the offer of oxygen and nutrients to the organs decreases, the consumption of oxygen and nutrients increases due to fever and immune reactions.

When the capillary system collapses, the organs and tissues suffer, and various forms of cell death in the organs begins including "programmed cell death" ("apoptosis"). This leads to organ damage, for example brain damage or kidney damage and ultimately to multiple organ dysfunction which is the direct cause of the patient dies.

Mild induced hypothermia (cooling to 32 0C-34 0C) affects at least 5 core areas in the pathophysiology of septic shock: 1) inhibition of inflammation 2) inhibition of apoptosis ("programmed cell death"), 3) antithrombotic, 4) decreases the metabolism and 5) inhibits bacterial growth and production of toxins.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 50 years of age.
2. Severe sepsis /septic shock = SIRS + suspected infection+hypotension Mean Arterial Blood Pressure (MAP) <70 mmHg,
3. Admitted to the participating intensive care units (ICU)
4. Indication for intubation
5. Possibility of inclusion within 6 hours after septic shock/severe sepsis is diagnosed in the ICU. Patients admitted with septic shock/severe sepsis should be included within 6 hours after admission. If a patient is not included within this period, that patient cannot be included within the same hospitalization.
6. The patient must have an expected stay in the ICU of more than 24 hours. Anticipated death within 24 hours after admission to the ICU does not exclude participation; however no decision of reduction of treatment level must have been taken. During this time period, probability that the patient is discharged to a floor department must not be likely (<10% probability).

Exclusion Criteria:

1. Patients are pregnant or breast feeding
2. The findings of the initial screening, shows that the patient has a bleeding disorder and/or the patient has an uncontrollable bleeding and /or surgery within the last 24 hours
3. Persons who are detained under the Act on the use of coercion in psychiatry

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  All cause

SECONDARY OUTCOMES:
Renal failure | 30 days
  RIFLE criteria (R+I+F) eGFR decrease (ml/min/1.73 m2) eGFR decrease to <60 ml/min/1,73)
  + derivatives of the above
Respiratory | 30 days
  Use of Mechanical Ventilation on day 4 No. of days where Mechanical Ventilation is used Delta PaO2/FiO2 ratio until day 4
  +Derivatives of the above
Circulatory breakdown/Septic Shock | Measure on day 4
  Delta MAP days 1-4 Inotropic Score day 1-4 Achieved discontinuation of inotropics on day 4
Cerebral dysfunction | Day 1-4
  Delta RASS 1-4 CAM-ICU: Days with positive CAM-ICU within 72 h after awakening MiniMentalState Examination (MMSE)
Hepatic Failure | Days 1-4
  Delta Bilirubin 1-4 Fraction of subjects with Bilirubin level >21 micromoles/L on day 4
Coagulatory Failure | Until Day 4/10
  Delta Platelets day 1-4 Delta INR days 1-4 (and factor 2/7/10) Delta APTT (days 1-4) Total consumption of SAG-M on days 1-10 Occurrence of Severe bleeding (surgery demanding or CT-verified, fresh upper or lower G-I bleeding) Thromboelastography
Duration of clinical infection | Days 1-4 + 1-30
  Delta C-reactive protein day 1-4 Achieved decrease in CRP >30 % from day 1-4 PCT decrease (Quantitative) day 1-10
Number of days Free of Organ failure | 30 days
  Number of days Free of Organ failure until day 30:
  Need for Mechanical ventilation, need for inotropic, RIFLE criteria positive, positive CAM-ICU days.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ulrik S Jensen, MD, PhD, Study Director — CHIP & PERSIMUNE, Rigshospitalet, University of Copenhagen
Locations (11):
- Cleveland Clinic - Outcomes Research, Cleveland, Ohio, United States
- Denmark (9):
  - Bispebjerg Hospital, Copenhagen, Capital Region
  - Jens Ulrik S. Jensen, Copenhagen, Capital Region
  - Gentofte Hospital, Gentofte Municipality, Capital Region
  - Herlev Hospital, Herlev, Capital Region
  - Nordsjællands Hospital, Hillerød, Hillerød, Capital Region
  - Aarhus University Hospital, Skejby, Aarhus, Jutland
  - Horsens Hospital, Horsens, Jutland
  - Køge Hospital, Køge, Region Sealand
  - Roskilde Hospital, Roskilde, Region Sealand
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The Steering Committee will share data after reviewing study propositions - this to assure quality

REFERENCES:
- [Derived] Itenov TS, Johansen ME, Bestle M, Thormar K, Hein L, Gyldensted L, Lindhardt A, Christensen H, Estrup S, Pedersen HP, Harmon M, Soni UK, Perez-Protto S, Wesche N, Skram U, Petersen JA, Mohr T, Waldau T, Poulsen LM, Strange D, Juffermans NP, Sessler DI, Tonnesen E, Moller K, Kristensen DK, Cozzi-Lepri A, Lundgren JD, Jensen JU; Cooling and Surviving Septic Shock (CASS) Trial Collaboration. Induced hypothermia in patients with septic shock and respiratory failure (CASS): a randomised, controlled, open-label trial. Lancet Respir Med. 2018 Mar;6(3):183-192. doi: 10.1016/S2213-2600(18)30004-3. Epub 2018 Jan 8. PMID 29325753
- [Derived] Johansen ME, Jensen JU, Bestle MH, Ostrowski SR, Thormar K, Christensen H, Pedersen HP, Poulsen L, Mohr T, Kjaer J, Cozzi-Lepri A, Moller K, Tonnesen E, Lundgren JD, Johansson PI. Mild induced hypothermia: effects on sepsis-related coagulopathy--results from a randomized controlled trial. Thromb Res. 2015 Jan;135(1):175-82. doi: 10.1016/j.thromres.2014.10.028. Epub 2014 Nov 5. PMID 25466837